CLINICAL TRIAL: NCT06806657
Title: A Phase 4 Open-label Study to Evaluate the Safety After Switching to CSL312 (Garadacimab) From Current Prophylactic HAE Treatment in Subjects With HAE ≥ 12 Years of Age
Brief Title: Safety Study in Subjects ≥ 12 Years of Age With Hereditary Angioedema Switching to Garadacimab
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSL312_4002; 2024-517757-27-00 (Other: EU CT Number)
Record Dates: First submitted 2025-02-03; First posted 2025-02-04 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Angioedema
Keywords: Autosomal dominant disease; Hereditary angioedema attack; Monoclonal antibody
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Garadacimab (Experimental)
  Interventions: Biological: Garadacimab

INTERVENTIONS:
Biological: Garadacimab — Participants will receive a loading dose of garadacimab, followed by once monthly garadacimab administration for 2 months. Garadacimab will be given as a subcutaneous injection. The timing for the administration of the loading dose (first administration of garadacimab) is determined by the dosing schedule of the current HAE prophylactic treatment. No washout necessary.
  Other Names: CSL312 and Factor XIIa inhibitor monoclonal antibody

SUMMARY:
This study is designed to evaluate the safety after switching to garadacimab from another prophylactic hereditary angioedema (HAE) treatment (marketed kallikrein [KK] inhibitor or plasma-derived C1-esterase inhibitor [pdC1INH]prophylactic) when administered once monthly for approximately 3 months in participants aged greater than or equal to (>=) 12 years with HAE.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 12 years at the time of providing written informed consent / assent.
* Have a history of response to on-demand HAE treatment for the treatment of acute HAE attacks.
* Documented laboratory diagnosis in medical records of C1-esterase inhibitor hereditary angioedema (HAE-C1INH) type 1 or type 2:

  * Documented clinical history consistent with HAE (subcutaneous or mucosal, nonpruritic swelling episodes without accompanying urticaria),
  * C1-esterase inhibitor (C1INH) antigen concentration or functional activity less than (<) 50% of normal as documented in the participant's medical record, or
  * C4-antigen concentration below the lower limit of the reference range as documented in the participant's medical record.

For HAE-nC1INH: Documented clinical history consistent with HAE (subcutaneous or mucosal, nonpruritic swelling episodes without accompanying urticaria); an HAE-associated FXII gene mutation (eg, FXII point mutation Thr328Lys or Thr328Arg, or deletion of 72 base pairs [c.971_1018 + 24del72], or duplication of 18 base pairs [c.892-909dup]), as documented in the participant's medical record, OR an HAE-associated plasminogen gene mutation (PLG) gene mutation (eg, PLG point mutation Lys330Glu), as documented in the participant's medical record; C1INH antigen concentration or functional activity 70 to 120% of the normal level, as documented in the participant's medical record.

• Use of lanadelumab, berotralstat, or pdC1INH for the prophylactic treatment of HAE and be on a stable (consistent) dose / regimen of such medication for at least 3 months prior to Screening.

Exclusion Criteria:

* Concomitant diagnosis of another form of angioedema, such as idiopathic or acquired angioedema or recurrent angioedema associated with urticaria.
* Use of androgens, antifibrinolytics, or investigational products (other than garadacimab) for routine prophylaxis against HAE attacks.
* Known or suspected hypersensitivity to monoclonal antibody therapy or hypersensitivity to the active substance (garadacimab) or to any of the excipients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to Day 95 (End of study [EoS])
Percentage of Participants With TEAEs | Up to Day 95 (EoS)
Number of TEAEs | Up to Day 95 (EoS)
Rate of TEAEs per injection | Up to Day 95 (EoS)
Rate of TEAEs per participant year | Up to Day 95 (EoS)

SECONDARY OUTCOMES:
Number of Participants With: Serious Adverse Events (SAEs), Deaths, Related TEAEs, TEAEs leading to study discontinuation, TEAEs by severity, Laboratory Findings Reported as an AE, and Adverse Events of Special Interest (AESI) | Up to Day 95 (EoS)
  The AESIs for garadacimab are severe hypersensitivity including anaphylaxis.
Percentage of Participants With: SAEs, Deaths, Treatment Related TEAEs, TEAEs leading to study discontinuation, TEAEs by severity, Laboratory Findings Reported as an AE, and AESI | Up to Day 95 (EoS)
Number of SAEs, Deaths, Treatment Related TEAEs, TEAEs leading to study discontinuation, TEAEs by severity, AESI and Laboratory Findings Reported as an AE, and AESI | Up to Day 95 (EoS)
Rate per injection of: SAEs, Deaths, Treatment Related TEAEs, TEAEs leading to study discontinuation, TEAEs by severity, Laboratory Findings Reported as an AE, and AESI | Up to Day 95 (EoS)
Rate per participant year of: SAEs, Deaths, Treatment Related TEAEs, TEAEs leading to study discontinuation, TEAEs by severity, Laboratory Findings Reported as an AE, and AESI | Up to Day 95 (EoS)
Number of Participants with Anti-garadacimab Antibodies | Up to Day 95 (EoS)
Percentage of Participants with Anti-garadacimab Antibodies | Up to Day 95 (EoS)
Plasma Concentrations of Garadacimab | Up to Day 95 (EoS)
Percentage of Participants who Indicated Their Preference for Garadacimab | Up to Day 95 (EoS)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (6):
- United States (5):
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Allergy and Asthma Clinic of Northwest Arkansas, Bentonville, Arkansas
  - Donald Levy M.D., Orange, California
  - Raffi Tachdjian MD, Inc., Santa Monica, California
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
- Clinique Spécialisée en Allergie de la Capitale, Québec, Canada

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (i.e. FDA, EMA) is complete and the primary publication is available
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.